CLINICAL TRIAL: NCT01354405
Title: The Effect of Lanreotide on Volume of Polycystic Liver and Kidney in Autosomal Dominant Polycystic Kidney Disease
Brief Title: Somatostatin Analogues as a Volume Reducing Treatment of Polycystic Livers (RESOLVE)
Acronym: RESOLVE
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: PCLD 10-03
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Polycystic Liver Disease
MeSH Terms: conditions — Polycystic liver disease | interventions — lanreotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lanreotide
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Lanreotide — 120 mg every 28 days intramuscular
  Other Names: Somatuline

SUMMARY:
The aim of this study is to determine the effect of Lanreotide on polycystic liver and kidneys in patients with autosomal dominant polycystic kidney disease.

DETAILED DESCRIPTION:
The aim of this single center observational study is to assess the effect of lanreotide on polycystic liver and kidney. This is achieved by assessing total liver and kidney volume, and several urinary markers that could predict kidney damage or kidney dysfunction, such as GFR, blood pressure, and urinary tubular damage markers and serum biomarker FGF23.

The investigators aim to include 43 patients affected by a polycystic liver due to ADPKD. The duration of the trial will be 28 weeks. The treatment will be 24 weeks and the first screening visit will take place four weeks before start of treatment. Eligible patients will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADPKD with polycystic liver (> 20 liver cysts)
* Renal function MDRD >40 ml/hr
* Informed consent, patients are willing and able to comply with the study drug regimen and all other study requirements

Exclusion Criteria:

* Kidney transplantation
* Renal failure requiring hemodialysis
* Use of oral contraceptives or estrogen suppletion
* Women who are pregnant or breastfeeding
* History of cardiac/pulmonary disease; symptomatic gallstones, pancreatitis, etc
* Intervention (aspiration or surgical intervention) within three months from baseline
* Treatment with somatostatin analogues within three months from baseline
* Mental illness that interferes with the patient ability to comply with the protocol
* Drug or alcohol abuse within one year from baseline
* Abnormal liver function tests, as determined by blood test (except isolated elevated GGT and AP, which occurs frequently in PLD)
* Clinical diagnosis of pancreatitis
* Diagnosis of diabetes mellitus, as determined by blood test and medical history
* Use of drugs that can interact with lanreotide, such as cyclosporin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ADPKD patients in Radboud University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Liver volume | 24 weeks
  Change in total liver volume between baseline and 24 weeks, as determined by CT volumetry

SECONDARY OUTCOMES:
Kidney volume | 24 weeks
  Change in kidney volume between baseline and 24 weeks, as determined by CT volumetry
Glomerular filtration rate | 24 weeks
  Change in GFR between baseline and 24 weeks, as determined by serum and 24 hrs urinary creatinine measurement
Urinary tubular damage markers | 24 weeks
  Change in urinary tubular damage markers between baseline and 24 weeks
Symptoms | 24 weeks
  Change in symptoms between baseline and 24 weeks, assessed by GI-questionnaire
Blood pressure | 24 weeks
  Change in blood pressure between baseline and 24 weeks
quality of life | 24 weeks
  Change in quality of life between baseline and 24 weeks, measured by EuroQoL-questionnaire
Adverse events | 24 weeks
  All adverse events that occur during 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joost PH Drenth, MD, PhD, Principal Investigator — Radboud University Hospital
Locations (1):
- Radboud University Hospital, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] van Keimpema L, Nevens F, Vanslembrouck R, van Oijen MG, Hoffmann AL, Dekker HM, de Man RA, Drenth JP. Lanreotide reduces the volume of polycystic liver: a randomized, double-blind, placebo-controlled trial. Gastroenterology. 2009 Nov;137(5):1661-8.e1-2. doi: 10.1053/j.gastro.2009.07.052. Epub 2009 Jul 29. PMID 19646443
- [Derived] Gevers TJ, Hol JC, Monshouwer R, Dekker HM, Wetzels JF, Drenth JP. Effect of lanreotide on polycystic liver and kidneys in autosomal dominant polycystic kidney disease: an observational trial. Liver Int. 2015 May;35(5):1607-14. doi: 10.1111/liv.12726. Epub 2014 Dec 1. PMID 25369108
- [Derived] Gevers TJ, Chrispijn M, Wetzels JF, Drenth JP. Rationale and design of the RESOLVE trial: lanreotide as a volume reducing treatment for polycystic livers in patients with autosomal dominant polycystic kidney disease. BMC Nephrol. 2012 Apr 4;13:17. doi: 10.1186/1471-2369-13-17. PMID 22475206